CLINICAL TRIAL: NCT00450749
Title: Phase II Placebo Controlled Trial of Preoperative Lycopene Supplementation in Prostate Cancer Patients
Brief Title: Lycopene in Treating Patients Undergoing Radical Prostatectomy for Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2009-00857; NCI-2009-00857 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MSKCC-06118; MDA-CC-2006-0388; CDR0000653464; CDR0000532938; 06-118; 2006-0388 (Other: M D Anderson Cancer Center); MDA04-3-01 (Other: DCP); P30CA016672 (NIH); N01CN35159 (NIH)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Results first posted 2012-07-16 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Adenocarcinoma of the Prostate; Stage I Prostate Cancer; Stage II Prostate Cancer; Stage III Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lycopene

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm I (placebo) (Placebo Comparator): Patients receive placebo PO QD for 4-7 weeks, and then undergo radical prostatectomy.
  Interventions: Other: placebo; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis
- Arm II (low-dose lycopene) (Experimental): Patients receive low-dose lycopene PO QD for 4-7 weeks, and then undergo radical prostatectomy.
  Interventions: Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis; Drug: lycopene
- Arm III (high-dose lycopene) (Experimental): Patients receive high-dose lycopene PO QD for 4-7 weeks, and then undergo radical prostatectomy.
  Interventions: Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis; Drug: lycopene

INTERVENTIONS:
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm I (placebo)
Procedure: therapeutic conventional surgery — Undergo radical prostatectomy
Other: laboratory biomarker analysis — Correlative studies
Drug: lycopene — Given PO
  Other Names: all-trans-Lycopene; Lyc-O-Mato; LYCO; psi,psi-Carotene
  Arms: Arm II (low-dose lycopene); Arm III (high-dose lycopene)

SUMMARY:
This randomized phase II trial studies how well different doses of lycopene work in treating patients undergoing radical prostatectomy for prostate cancer. The use of lycopene, a substance found in tomatoes, may keep prostate cancer from growing or coming back after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the differences in tissue concentrations of lycopene in patients with prostate cancer undergoing radical prostatectomy treated with different doses of neoadjuvant lycopene supplementation.

II. Compare the change in serum lycopene concentration from baseline and at 4-7 weeks in patients treated with different doses of lycopene.

SECONDARY OBJECTIVES:

I. Determine the effect of this treatment in down-regulating 5-alpha-reductase activity by measuring the change in the ratio of testosterone (T) to dihydrotestosterone (DHT) in serum at baseline and at 4-7 weeks and the ratio of T:DHT in prostatic surgical tissue post-treatment.

II. Determine the effect of this treatment in attenuating baseline blood serum concentrations of total prostate-specific antigen (PSA), free PSA, and human kallikrein 2 in these patients.

III. Determine the effect of this treatment on growth potential by examining post-treatment radical prostatectomy tissue specimens for proliferative index (PI) by Ki-67 expression, apoptotic index (AI) by TUNEL assay, and PI:AI ratio in these patients.

IV. Determine the effect of this treatment in modulating putative biomarkers of lycopene efficacy, including serum concentrations of insulin-like growth factor (IGF)-1 and IGF binding protein-3, lymphocyte oxidative DNA damage capacity by Comet assay, and GST-pi expression in prostatic tissue from these patients.

V. Compare the histological effect of different doses of lycopene on putative prognostic features, including the presence and extent of high-grade prostatic intraepithelial neoplasia, prostatitis, total tumor volume, local invasion (vascular and lymphatic, capsular, seminal vesicle), pathologic stage, Gleason score, surgical margins, and lymph node status in these patients.

VI. Determine the effect of this treatment in modulating the RNA expression of androgen-related genes by microarray analysis in these patients.

OUTLINE:

This is a randomized, placebo-controlled, double-blind, multicenter study. Patients are stratified according to participating center. Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive placebo orally (PO) once daily (QD) for 4-7 weeks, and then undergo radical prostatectomy.

ARM II: Patients receive low-dose lycopene PO QD for 4-7 weeks, and then undergo radical prostatectomy.

ARM III: Patients receive high-dose lycopene PO QD for 4-7 weeks, and then undergo radical prostatectomy.

Tumor samples are collected from prostatectomy for laboratory studies, including GST-pi expression by immunohistochemistry; histological analysis; microarray analysis of androgen-related genes; ratio of testosterone (T) to dihydrotestosterone (DHT); Ki-67 expression; and lycopene tumor-concentration measurement.

Patients undergo blood collection at baseline, week 4, and week 7 for laboratory studies, including serum lycopene concentration measurement; level of T or DHT by high-performance liquid chromatography/tandem mass spectrometry (HPLC/MS/MS) analysis; serum concentrations of total prostate-specific antigen (PSA), free PSA, and human kallikrein 2; lymphocyte oxidative DNA damage capacity; and serum concentrations of insulin-like growth factor (IGF)-1 and IGF binding protein-3 by radioimmunological assay.

ELIGIBILITY:
Criteria:

* Creatinine normal
* Biopsy-confirmed adenocarcinoma of the prostate
* Localized disease
* Planned radical prostatectomy
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* WBC >= 3,000/mm^3
* Platelet count >= 100,000/mm^3
* Bilirubin normal
* AST and ALT =< 2.5 times upper limit of normal
* Fertile patients must use effective barrier contraception
* No other invasive cancer (except nonmelanoma skin cancer) within the past 2 years
* Patients who received curative treatment and have shown no evidence of recurrence within the past 2 years are eligible
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to lycopene (e.g., other carotenoids, including lutein and beta-carotene)
* More than 30 days since prior regular (> once weekly) lycopene supplementation (>= 15 mg/day) and meets the following criteria: no more than 2 servings of tomato sauce, juice, or soup per week; no more than 4 servings of grapefruit, raw tomato, or watermelon per week
* Must not consume 1 serving of tomato sauce, juice, or soup per week AND more than 2 servings of grapefruit, raw tomato, or watermelon per week
* More than 30 days since prior and no concurrent investigational medication
* No concurrent chemotherapy, radiotherapy, hormonal therapy, or immunotherapy
* No history of allergy to foods containing lycopene (e.g., tomatoes or tomato products, watermelon, guava, and pink grapefruit)
* No concurrent uncontrolled illness including, but not limited to, any of the following: ongoing or active infection; symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia; psychiatric illness/social situations that would limit compliance with study requirements
* No prior therapy for prostate cancer, including radiotherapy to the prostate or pelvis, androgen ablation, or antiandrogen systemic therapy
* No other concurrent lycopene (>= 15 mg/day)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Eastham, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 11, 2008 to April 15, 2009. All recruitment was done in a medical clinic setting, and all participants enrolled at Memorial Sloan-Kettering Cancer Center.
Pre-assignment Details: There were eleven participants registered, one participant was excluded from the trial before assignment to groups making only ten randomized.
Groups:
- Arm I Placebo: Placebo once daily for 4-7 weeks.
- Arm II Low Dose Lycopene: 30 mg/day oral Lycopene for 4-7 weeks.
- Arm III High-Dose Lycopene: 60 mg/day oral Lycopene for 4-7 weeks.
Period: Overall Study
Arm/Group | Arm I Placebo | Arm II Low Dose Lycopene | Arm III High-Dose Lycopene
Started | 3 | 3 | 4
Completed | 3 | 2 | 2
Not Completed | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Noncompliant | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I Placebo | Arm II Low Dose Lycopene | Arm III High-Dose Lycopene | Total
Number analyzed (Participants) | 3 | 3 | 4 | 10
Age, Continuous [Median (Full Range); unit: years] | 71 [56 to 72] | 56 [45 to 71] | 66 [52 to 68] | 66.5 [45 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 3 | 3 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Lycopene in Prostatic Surgical Tissue
Description: Total tissue lycopene concentrations in radical prostatectomy specimens in participants receiving 6 weeks (± 1 week) of preoperative supplementation with 60 mg/day lycopene, 30 mg/day lycopene, or placebo. Concentration of lycopene in prostatic surgical tissue calculated using the high-performance liquid chromatography (HPLC) method.
Time Frame: At 4-7 weeks
Population: Tissue samples collected from five participants for measurement of lycopene levels, representing only 50% (5 of 10) of the participants' enrolled on-trial.
Measure: Number; unit: ug/dL
Arm/Group | Arm I Placebo | Arm II Low Dose Lycopene | Arm III High-Dose Lycopene
Number analyzed (Participants) | 2 | 2 | 2
ug/dL
  Sample 1 | 0.663 | 0.378 | 0.723
  Sample 2 | 0.165 | 0.749 | NA — A second tissue sample was not collected.

2. Primary Outcome: Serum Levels (ug/dL) of Total Lycopene at Baseline and During Treatment by Group
Description: Serum levels (ug/dL) of total lycopene at baseline and during treatment by group were measured.
Time Frame: Baseline and weeks 4 and 7
Population: 10 participants were analyzed at Baseline versus 8 at Week 4 and versus 5 at Week 7 due to drop out rate.
Measure: Median (Full Range); unit: ug/dL
Arm/Group | Arm I Placebo | Arm II Low Dose Lycopene | Arm III High-Dose Lycopene
Number analyzed (Participants) | 3 | 3 | 4
ug/dL
  Baseline | 25.3 [16.2 to 38.9] | 32.0 [31.1 to 99.0] | 22.7 [21.2 to 24.2]
  Week4: number analyzed (Participants) | 3 | 2 | 3
  Week4 | 98.7 [77.4 to 127.7] | 40.4 [18.7 to 62.1] | 61.5 [42.7 to 86.3]
  Week 7: number analyzed (Participants) | 1 | 2 | 2
  Week 7 | 125.8 [125.8 to 125.8] | 52.8 [24.7 to 81.0] | 44.4 [39.6 to 49.2]

3. Secondary Outcome: Ratio of T:DHT in Prostatic Surgical Tissue
Time Frame: At 4-7 weeks
Population: Because the trial closed before the accrual goals were met, therefore only the primary measures were analyzed. No secondary analyses were done.
Arm/Group | Arm I Placebo | Arm II Low Dose Lycopene | Arm III High-Dose Lycopene
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Serum Concentrations of Total Prostate-specific Antigen (PSA), Free PSA, and Human Kallikrein 2
Time Frame: Baseline and at 4-7 weeks
Population: as for outcome 3
Arm/Group | Arm I Placebo | Arm II Low Dose Lycopene | Arm III High-Dose Lycopene
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Growth Potential Assessed by the Ratio of Proliferation (Ki-67):Apoptosis (TUNEL) in Prostatic Surgical Tissue
Time Frame: At 4-7 weeks
Population: as for outcome 3
Arm/Group | Arm I Placebo | Arm II Low Dose Lycopene | Arm III High-Dose Lycopene
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Serum Concentrations of Insulin-like Growth Factor (IGF)-1 and IGF Binding Protein-3
Time Frame: At baseline and at 4-7 weeks
Population: as for outcome 3
Arm/Group | Arm I Placebo | Arm II Low Dose Lycopene | Arm III High-Dose Lycopene
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Lymphocyte Oxidative DNA Damage Capacity as Measured by Comet Assay
Time Frame: At baseline and at 4-7 weeks
Population: as for outcome 3
Arm/Group | Arm I Placebo | Arm II Low Dose Lycopene | Arm III High-Dose Lycopene
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Expression of GST-pi in Prostatic Surgical Tissue
Time Frame: At 4-7 weeks
Population: as for outcome 3
Arm/Group | Arm I Placebo | Arm II Low Dose Lycopene | Arm III High-Dose Lycopene
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Histological Characteristics of Prostatic Surgical Tissue
Time Frame: At 4-7 weeks
Population: as for outcome 3
Arm/Group | Arm I Placebo | Arm II Low Dose Lycopene | Arm III High-Dose Lycopene
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Modulation of Expression of Androgen-related Genes as Measured by Microarray in Prostatic Surgical Tissue
Time Frame: At 4-7 weeks
Population: as for outcome 3
Arm/Group | Arm I Placebo | Arm II Low Dose Lycopene | Arm III High-Dose Lycopene
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Ratio of Testosterone (T) to Dihydrotestosterone (DHT) in Serum
Time Frame: Baseline and at 4-7 weeks
Population: as for outcome 3
Arm/Group | Arm I Placebo | Arm II Low Dose Lycopene | Arm III High-Dose Lycopene
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 13 months
Arm/Group | Arm I Placebo | Arm II Low Dose Lycopene | Arm III High-Dose Lycopene
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I Placebo (N=3) | Arm II Low Dose Lycopene (N=3) | Arm III High-Dose Lycopene (N=4)
Dizziness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (General disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cardia Arrythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less